CLINICAL TRIAL: NCT01271088
Title: Phase 3 Study of Protective Effect of N-acetylcysteine Against From Ototoxicity
Brief Title: Protective Effect of N-acetylcysteine Against From Ototoxicity
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ismail Kocyigit, TC Erciyes University Department of Nephrology, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EUTF 2010/32
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2011-11-16 (Estimated); Status verified 2011-11

CONDITIONS: Hearing Loss, Extreme
Keywords: ototoxicity; aminoglycoside; vancomycine; peritoneal dialysis; peritonitis
MeSH Terms: conditions — Deafness; Ototoxicity; Peritonitis | interventions — Acetylcysteine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N-acetylcysteine (Experimental): N-acetylcysteine: Experimental N-acetylcysteine 600 mg twice daily + vancomycine and/or amikacin
  Interventions: Drug: N-acetylcysteine
- Control (No Intervention): Vancomycine and/or amikacin alone
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — N-acetylcysteine 600 mg twice a day,one week after administration of antibiotics
  Other Names: NAC

SUMMARY:
Peritonitis is currently one of the leading complications of continuous ambulatory peritoneal dialysis (CAPD). Aminoglycosides and vancomycin are used in the treatment of CAPD peritonitis despite their potential risk for ototoxicity. NAC is a molecule used in the treatment and prophylaxis of many diseases related to oxidative stress. The aim of this study was to examine whether ototoxicity due to antibiotics used in the treatment of CAPD peritonitis can be prevented by N-acetylcysteine

DETAILED DESCRIPTION:
NAC, a thiol-containing antioxidant because of this,we want to investigate antioxidant status.

ELIGIBILITY:
Inclusion Criteria:

* End-stage renal disease
* Undergoing continuous ambulatory peritoneal dialysis as a renal replacement therapy
* Developing the first continuous ambulatory peritoneal dialysis related peritonitis episode

Exclusion Criteria:

* Being treated with aminoglycoside antibiotics and vancomycine within the previous 3 months
* Detection of mechanical occlusion of external ear
* Having signs of disturbed integrity of tympanic membrane on otoscopy or tympanometry
* History of a continuous ambulatory peritoneal dialysis related peritonitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Threshold hearing levels | 4 weeks
  Ototoxicity was defined as an increase in the auditory threshold by at least 20 dB at any one test frequency, or at least 10 dB at any two adjacent frequencies, or loss of response at three consecutive frequencies between the baseline and follow-up studies in the worse ear.

CONTACTS AND LOCATIONS:
Overall Officials: Ismail Kocyigit, MD, Principal Investigator — TC Erciyes University
Locations (1):
- Erciyes University, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Kocyigit I, Vural A, Unal A, Sipahioglu MH, Yucel HE, Aydemir S, Yazici C, Ilhan Sahin M, Oymak O, Tokgoz B. Preventing amikacin related ototoxicity with N-acetylcysteine in patients undergoing peritoneal dialysis. Eur Arch Otorhinolaryngol. 2015 Oct;272(10):2611-20. doi: 10.1007/s00405-014-3207-z. Epub 2014 Jul 30. PMID 25073872